CLINICAL TRIAL: NCT01567410
Title: Randomized Controlled Trial to Evaluate the Effect of E-learning on Nurses Ability to Assess Patient Risk for Pressure Ulcers and Pressure Ulcer Classification
Brief Title: Evaluation of an E-learning Program for Assessing Pressure Ulcer Risk and Pressure Ulcer Classification - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sophies Minde Ortopedi (Industry); Norwegian Nurses Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 2012/471
Record Dates: First submitted 2012-03-20; First posted 2012-03-30 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Learning; Efficiency
Keywords: e-learning; education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional Classroom training (Other): one group of nurses receive traditional classroom training to learn about the braden scale and pressure ulcer classification
  Interventions: Other: traditional classroom training
- e-learning (Other): one group of nurses receive e-learning as a training method to learn about the braden scale and classification of pressure ulcer
  Interventions: Other: e-learning

INTERVENTIONS:
Other: e-learning — Braden scale and pressure ulcer classification
  Arms: e-learning
Other: traditional classroom training — Braden scale and pressure ulcer classification
  Arms: traditional Classroom training

SUMMARY:
The purpose of this study is to determine wether e-learning is a more effective than traditional classroom teaching at norwegian nurses ability to use the Braden risk assessment scale and pressure ulcer classification.

DETAILED DESCRIPTION:
Most pressure ulcers (PU)can be prevented and assessment of the patient skin and risk factors for pressure ulcers is the first step. Epidemiological studies are also an important element in the prevention of PU and requires consistent registration based on standardized definitions and tools. Staff knowledge is critical in this work. However showed a Norwegian pilot study on the prevalence of PU deficient knowledge among nursing staff in terms reliable classification of PU and PU-assessment of risk. The pilot study showed the need for training to reduce the incidence of pressure ulcers and to ensure data quality in future studies.

E-learning is an alternative to traditional courses and will help to streamline and standardize training by allowing a larger number of personnel be reached with this method of training. It is not designed Norwegian e-learning program that addresses the use of risk assessment instrument or classification of PU. We have developed one program to train personnel in the PU-classification and risk assessment and plan to evaluate this. The program will be an important contribution to the PU-prevention as well as the program will be used in the execution of a multicenter prevalence study of PU-prevalence.

Nurses will randomly assign to a lecture, e-learning or to a control group. The lecture and e-learning are based on the same content. The nurses will score five patient cases with braden scale before and after intervention and 20 pictures of pressure ulcers in different categories before and 40 after intervention. The control group will only do a pretest.

ELIGIBILITY:
Inclusion Criteria:

* registered nurse and postgraduate nurse working at somatic ward, emergency ward, surgical department, intensive care unit,recovery, nursinghome or homecare

Exclusion Criteria:

* working at maternity ward, pediatric ward, psychiatric ward

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Braden scale score | up to 24 weeks
  Both subscale and total sum on five patient cases are collected using Braden scale at baseline (right before and right after the intervention) to see if the intervention is giving a change in the score. At 12 weeks and 24 weeks to see if the knowledge remains.

SECONDARY OUTCOMES:
Pressure ulcer classification | up to 24 weeks
  pressure ulcer photos in different categories are scored by normal skin, category 1,2, 3 or 4. Baseline (right before and right after the intervention) to see if the intervention is giving a change in the score. At 12 weeks and 24 weeks to see if the knowledge remains.

CONTACTS AND LOCATIONS:
Overall Officials: Ida M. Bredesen, PhDcandidate, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Norway